CLINICAL TRIAL: NCT04200391
Title: Glucagon Response in Patients With Type 1 Diabetes Mellitus Following a Very Low Carbohydrate
Brief Title: Very Low Carbohydrate Diets and Glucagon Response in T1DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Belinda Lennerz, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00030039_3
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Type1diabetes
Keywords: nutrition; very low carbohydrate diet; ketogenic diet; nutritional ketosis; glucagon; hypoglycemia; glycogen; ketosis; ketones
MeSH Terms: conditions — Hypoglycemia; Ketosis

STUDY DESIGN:
Intervention Model Description: Participants will receive a very low carbohydrate diet for 12 weeks and undergo a glucagon challenge during weeks 5-12 to assess glycemic response.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very low carbohydrate diet (Experimental): Dietary Intervention, food delivery
  Interventions: Other: Very low carbohydrate diet

INTERVENTIONS:
Other: Very low carbohydrate diet — All meals will be delivered and participants will consume study foods exclusively. Participants will receive a fiber supplement with each meal as needed to promote digestive health, and a daily multi-vitamin, magnesium and omega-3 supplement to ascertain micronutrient sufficiency. Participants will be weighed at each study visit and the diet plan will be adjusted for satiety and weight-maintenance.
  The diet composition will be as follows: 5% carbohydrate, 75% fat, 20% protein.

SUMMARY:
Despite major technological advances, management of type one diabetes mellitus (T1D) remains suboptimal, putting millions of people at risk for immediate and long-term complications. After meals, a mismatch between carbohydrate absorption rate and insulin action typically leads to alternating periods of hyper- and hypoglycemia. A conceptually promising approach to control both problems is dietary carbohydrate restriction to reduce postprandial blood glucose changes and insulin needs. In a prior survey study, the investigators documented exceptional glycemic control (HbA1c 5.67%) and low acute complication rates among 316 children and adults with T1D consuming a very-low-carbohydrate (VLC) diet. Despite these promising preliminary results, the use of VLC diets for T1D remain controversial, because of their restrictive nature and theoretical concerns regarding growth, ketoacidosis and hypoglycemia risks and efficiency of glucagon treatment for hypoglycemia. Glucagon is used as a rescue medication during severe hypoglycemia and increases blood glucose levels by mobilizing liver glycogen stores. If these stores are depleted during carbohydrate restriction, glucagon response may be inadequate and put individuals at risk for refractory hypoglycemia. A physiologic study has shown a blunted but still adequate response to glucagon in n=10 participants after following a VLCD for 1 week. Longer-term studies have not been done.

To test the hypotheses that glucagon response remains adequate while following a VLC diet in the longer term, the investigators will conduct a glucagon challenge in participants who are assigned to the VLC arm of a randomized-controlled feeding study in 32 young adults with T1D who will receive a VLC vs a standard diet for 12 weeks. After an overnight fast, twelve participants in the VLC arm will receive IV insulin to lower blood glucose levels to 60 mg/dL, followed by a glucagon injection and monitoring of blood glucose levels and other metabolic fuels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with T1D for at least 1 year
* Age 18 to 40 years
* Tanner stage ≥ IV
* BMI 18.5-35 kg/m2
* Stable glycemic control (HbA1c 6.5-9%)
* Use of a continuous glucose monitor (CGM)
* Use of an insulin pump
* Attendance of at least 1 diabetes care visit over the past 12 months (including virtual)

Exclusion Criteria:

* Ketoacidosis or severe hypoglycemia with seizure or coma in the past 6 months
* Dietary restrictions or intolerances that are incompatible with the planned food deliveries, e.g. celiac disease, gastroparesis, certain food allergies
* Following a weight-loss or otherwise restrictive diet
* Vigorous exercise >2 hours on >3 days a week
* History of an eating disorder or at risk for eating disorder, assessed by the Eating Disorders Diagnostic Scale (EDDS)
* Major medical illness or use of medications other than insulin and metformin that could interfere with metabolic or glycemic variables
* Significant psychiatric illness
* Smoking, use of recreational drugs, or excessive alcohol consumption
* Pregnancy or breastfeeding
* Anemia
* For participants who undergo MRI:

  1. Standard MRI exclusion criteria
  2. Irregular menses
  3. Use of psychotropic medication other than SSRIs or other mild antidepressant or anxiety medications (unless these medications are safe to be held for several days to allow for the acquisition of MRI data).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Glucagon treatment success, defined as an increase in glucose level to ≥ 70 mg/dL or an Increase of ≥ 20 mg/dL from glucose nadir within 30 minutes after receiving 1 mg glucagon IM | week 5-12 on the very low carbohydrate diet
  Point-of-care blood glucose levels will be measured pre-dose and every 5 minutes for 30 minutes and until BG is ≥ 70 mg/dL (whichever occurs later), then gradually spaced per MD orders to align with the rest of the labs

SECONDARY OUTCOMES:
Recovery from symptoms of hypoglycemia | week 5-12 on the very low carbohydrate diet
  Recovery from hypoglycemia symptoms will be assessed using a Hypoglycemia Symptoms Scale at baseline, when blood glucose is < 75 mg/dL, pre-dose, and at 15, 30, 45, 60, 75, and 90 minutes following administration of glucagon. The Hypoglycemia Symptoms Scale measures the intensity of 14 commonly experienced hypoglycemic symptoms on a scale from 0 (not present) to 6 (very intense). The higher the score, the more intense the hypoglycemia symptoms. The sum of each symptom score would yield a range of 0 to 84 (e.g., 14 x 6 = 84). The total score will be calculated as the sum of each symptom score and summarized at each time point.
Time to achieve glucagon treatment success | week 5-12 on the very low carbohydrate diet
  The mean time from glucagon administration to blood glucose ≥ 70 mg/dL or an increase ≥ 20 mg/dL in blood glucose from nadir. Point-of-care blood glucose levels will be measured pre-dose and every 5 minutes for 30 minutes and until BG is ≥ 70 mg/dL (whichever occurs later), then gradually spaced per MD orders to align with the rest of the labs.
Plasma levels of beta-hydroxybutyrate following glucagon administration | week 5-12 on the very low carbohydrate diet
  Levels will be measured at baseline, pre-dose, and at 10, 20, 30, 45, 60, and 90 minutes. Average levels at each time point, peak level, and area under the curve (AUC) will be reported.
Plasma levels of free fatty acids following glucagon administration | week 5-12 on the very low carbohydrate diet
  Levels will be measured at baseline, pre-dose, 10, 20, 30, 45, 60, and 90 minutes. Average levels at each time point, peak level, and area under the curve (AUC) will be reported.
Plasma glucose levels following glucagon administration | week 5-12 on the very low carbohydrate diet
  Levels will be measured at baseline, pre-dose, and at 10, 20, 30, 45, 60, and 90 minutes. Average levels at each time point, peak level, and area under the curve (AUC) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda S Lennerz, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided